CLINICAL TRIAL: NCT06180096
Title: Single Dose Oral Bioequivalence Study of Riociguat 2.5 mg Film Coated Tablets and 'Adempas' (Riociguat) 2.5 mg Filmtabletten (Film Coated Tablets) in Healthy Adult Male Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Riociguat 2.5 mg Film Coated Tablets and Adempas (Riociguat) 2.5 mg Film Coated Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1B02230
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riociguat film coated tablets (Experimental): Riociguat 2.5 mg film coated tablets
  Interventions: Drug: Riociguat film coated tablets; Drug: Adempas Filmtabletten
- Adempas Filmtabletten (Active Comparator): Adempas (Riociguat) 2.5 mg Filmtabletten
  Interventions: Drug: Riociguat film coated tablets; Drug: Adempas Filmtabletten

INTERVENTIONS:
Drug: Riociguat film coated tablets — 1 tablet of 2.5 mg Riociguat
Drug: Adempas Filmtabletten — 1 tablet of 2.5 mg Riociguat

SUMMARY:
Single dose oral bioequivalence study of Riociguat 2.5 mg film coated tablets and 'Adempas' (Riociguat) 2.5 mg Filmtabletten (film coated tablets) in healthy adult male subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers must fulfill all of the following inclusion criteria to be eligible for participation
2. in the study, unless otherwise specified. 1) Age: 18 to 45 years old, both inclusive. 2) Gender: Male
3. BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value should be rounded off to one
4. significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while
5. 18.45 rounds up to 18.5).
6. Able to communicate effectively with study personnel.
7. Willing to provide written informed consent to participate in the study.
8. Non-smokers and non-tobacco users (i.e. having no past history of smoking and
9. tobacco consuming for at least one year prior to study).
10. Volunteer must have sitting systolic blood pressure at least 100 mmHg and sitting
11. diastolic blood pressure at least 60 mmHg during screening.
12. Volunteer must agree to either abstain from sexual intercourse or use an acceptable
13. method of birth control from screening until 4 weeks after the last study procedure.
14. All volunteers must be judged by the principal or sub-investigator or physician as
15. normal and healthy during a pre-study safety assessment performed within 28 days of
16. the first dose of study medication which will include:

    1. A physical examination (clinical examination) with no clinically significant finding.
    2. Results within normal limits or clinically non-significant for the following tests: Hematology, Biochemistry, Urinalysis, Immunological Tests Additional tests and/or examinations (apart from mentioned in protocol) may be performed, if necessary, based on principal investigator discretion. All results will be assessed against the current laboratory normal ranges at the time of testing and a copy of the normal ranges used will be included in the study documentation.

       Exclusion Criteria:

       Volunteers must not be enrolled in the study if they meet any one of the following criteria:
       1. History of allergic responses to Riociguat or other related drugs, or any of its formulation ingredients.
       2. Have significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG recording].
       3. Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
       4. History or presence of bronchial asthma.
       5. Use of any hormone replacement therapy within 3 months prior to the first dose of study medication.
       6. A depot injection or implant of any drug within 3 months prior to the first dose of study medication.
       7. Use of CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see https://drug-interactions.medicine.iu.edu/MainTable.aspx).
       8. History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
       9. History of difficulty with donating blood or difficulty in accessibility of veins.
       10. A positive hepatitis screen (includes subtypes B & C).
       11. A positive test result for HIV antibody.
       12. Volunteers who have received a known investigational drug within seven elimination half-life of the administered drug prior to the first dose of study medication.
       13. Volunteers who have donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever is greater.
       14. History of difficulty in swallowing or of any gastrointestinal disease, which could affect drug absorption.
       15. Intolerance to venipuncture
       16. Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.
       17. Institutionalized volunteers.
       18. Use of any prescribed medications [including PDE5 inhibitors (such as sildenafil, tadalafil, vardenafil, nitrates or nitric oxide donors (such as amyl nitrite), soluble guanylate cyclase stimulators] within 14 days prior to the first dose of study medication.
       19. Use of any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
       20. Use of grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
       21. Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeinecontaining sodas, colas, etc.), recreational drugs (including poppers), alcohol or other alcohol containing products within 120 hours prior to the first dose of study medication.
       22. Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
       23. Volunteer having serum creatinine higher than upper limit of normal range in screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Maximum concentration obtained (Cmax) | 48 hours
  Two-sided 90% confidence interval for the test to reference ration of the population means is within 80.00% to 125.00% for each of the Ln-transformed data Cmax
AUC from time 0 to last collection time t (AUC) | 48 hours
  Two-sided 90% confidence interval for the test to reference ration of the population means is within 80.00% to 125.00% for each of the Ln-transformed data AUC0-t

SECONDARY OUTCOMES:
AUC from time 0 to infinity (AUC0-inf) | 48 hours
  Descriptive statistics
Time to reach maximum concentration Cmax (Tmax) | 48 hours
  Descriptive statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No